CLINICAL TRIAL: NCT01977040
Title: Optimal Management of Vasa Previa: Screening, Diagnosis and Management - A Retrospective Study.
Brief Title: Optimal Management of Vasa Previa Study - A Retrospective Study
Acronym: VasaPrevia
Status: Completed | Type: Observational
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Other Study IDs: OBX0025
Record Dates: First submitted 2013-10-04; First posted 2013-11-06 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Vasa Previa
Keywords: Vasa Previa
MeSH Terms: conditions — Vasa Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vasa Previa: Women with the diagnosis of Vasa Previa made during the pregnancy or at time of delivery who delivered between January 1, 2000 and December 31, 2012.

SUMMARY:
This is a multicenter retrospective observational study of women diagnosed with a vasa previa during pregnancy or at delivery who delivered between 2000 and 2012. The study hopes to be able to describe techniques utilized to screen for and diagnose vasa previa as well as to describe the maternal characteristics and identify potential underlying risk factors that may provide a basis for future screening recommendations for vasa previa and treatment protocols.

DETAILED DESCRIPTION:
This is a multicenter retrospective study of women identified as having a vasa previa during pregnancy or at the time of delivery who delivered between January 1, 2000 and December 31, 2012 at participating centers. The primary objective of the study is to describe techniques utilized to screen for and diagnose vasa previa.

* In those cases that were diagnosed antenatally, to describe the different management protocols utilized, correlate these management protocols with neonatal outcomes and support the management protocol that offers optimal outcomes for both mother and neonate.
* In those cases that were not diagnosed antenatally, to describe the clinical scenario surrounding delivery and the neonatal outcomes. Review the ultrasound reports and maternal characteristics to identify any potential risk factors for vasa previa that could have been identified antenatally in attempt to improve neonatal outcomes in the future.
* In all cases of diagnosed vasa previa (those diagnosed antepartum, intrapartum, and postpartum), to describe the maternal characteristics and identify potential underlying risk factors that may provide a basis for future screening recommendations and protocols. Due to the rarity of this diagnosis, the study hopes to include 100-250 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosed of vasa previa made either during the pregnancy via ultrasound or at time of delivery via clinical and/or pathologic investigation.
* Patient delivered between January 2000 through December 2012

Exclusion Criteria:

* No diagnosis or confirmation of vasa previa
* Delivered either before January 1, 2000 or after December 31, 2012

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women at participating site who have been identified as having a vasa previa between January 1, 2000 and December 31, 2012.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Garite, MD, Principal Investigator — Pediatrix Medical Group, Inc.
Locations (9):
- United States (9):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Good Samaritan Hospital, San Jose, California
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Saint Luke's Hospital, Kansas City, Kansas City, Missouri
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In a retrospective manner, we recruited all pregnancies complicated by vasa previa that delivery between January 1, 2000 and December 31, 2012 at nine Maternal Fetal Medicine Practices. The diagnosis of vasa previa was made either during the antenatal period by an ultrasound or at the time of delivery via clinical and/or pathologic investigation
Period: Overall Study
Arm/Group | Vasa Previa
Started | 68
Completed | 66
Not Completed | 2
Not completed — Vasa previa not confirmed | 2

BASELINE CHARACTERISTICS:
Population: Women with the diagnosis of Vasa Previa made during the pregnancy or at time of delivery who delivered between January 1, 2000 and December 31, 2012.
Arm/Group | Vasa Previa
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 0
Region of Enrollment [Number; unit: participants] — Enrolled in the US mostly western United States
  participants
    United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Profile of Techniques Utilized to Screen for and Diagnose Vasa Previa During Pregnancy.
Description: The primary outcome of the study it to describe antenatal techniques utilized to screen for and diagnose vasa previa. Vasa previa is when unprotected blood vessels implanted in the membranes or sac run from the placenta across the inside of the woman's cervix. Antepartum ultrasounds were conducted according to standard of care. Here we report the count of participants who were diagnosed during routine ultrasound exam. After initial diagnosis by ultrasound, Vasa Previa's were followed up by routine ultrasounds for confirmation prior to delivery.
Time Frame: Participants will be followed from time of diagnosis of vasa previa until the baby is born, an expected time frame of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vasa Previa
Number analyzed (Participants) | 66
Participants
  Antepartum Ultrasound, confirmed at delivery | 47
  Antepartum Ultrasound, not confirmed at delivery | 13
  Antepartum Ultrasound, resolved prior to delivery | 4
  No antepartum diagnosis, Vasa Previa at birth | 2

2. Primary Outcome: Gestational Age at Time of Diagnosis Stratified by Diagnostic Profile.
Time Frame: Participants will be followed from time of diagnosis of vasa previa during the second trimester up until delivery.
Population: Only 64 participants had vasa previa diagnosed via ultrasound during the antenatal period.
Measure: Mean (Full Range); unit: weeks
Arm/Group | Vasa Previa
Number analyzed (Participants) | 64
weeks
  Antepartum Ultrasound, confirmed at delivery: number analyzed (Participants) | 47
  Antepartum Ultrasound, confirmed at delivery | 27.0 [16 to 40]
  Antepartum Ultrasound, not confirmed at delivery: number analyzed (Participants) | 13
  Antepartum Ultrasound, not confirmed at delivery | 27.8 [16 to 32]
  Antepartum Ultrasound, resolved prior to delivery: number analyzed (Participants) | 4
  Antepartum Ultrasound, resolved prior to delivery | 19.8 [18 to 21]

3. Primary Outcome: Mode of Delivery Stratified by Diagnostic Profile.
Description: Mode of delivery (C/S - emergent, non-emergent, vaginal) stratified by diagnostic profile
Time Frame: At birth.
Measure: Count of Participants; unit: Participants
Groups:
- Emergent Cesarean Section: Cesarean Section prompted by a medical emergency.
- Non-Emergent Cesarean Section: Cesarean Section planned or non-emergency related.
- Vaginal Delivery: Delivered vaginally.
Arm/Group | Emergent Cesarean Section | Non-Emergent Cesarean Section | Vaginal Delivery
Number analyzed (Participants) | 10 | 51 | 5
Participants
  Antepartum Ultrasound, confirmed at delivery | 7 | 40 | 2
  Antepartum Ultrasound, not confirmed at delivery | 2 | 9 | 2
  Antepartum Ultrasound, resolved prior to delivery | 0 | 1 | 1
  No antepartum diagnosis, Vasa Previa at birth | 1 | 1 | 0

4. Primary Outcome: Gestational Age of Infant at Birth
Description: Gestational age of the infant noted in weeks at the time of birth
Time Frame: At birth.
Population: Mean Gestational age at delivery as well as Mean Gestational Age for those patients who delivered emergently and non-emergent are presented.
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Non-Emergent Cesarean Section and Vaginal Delivery: Cesarean Section planned or non-emergency related and Vaginal Deliveries were included in this data
Arm/Group | Emergent Cesarean Section | Non-Emergent Cesarean Section and Vaginal Delivery
Number analyzed (Participants) | 10 | 56
weeks
  Antepartum Ultrasound, confirmed at delivery: number analyzed (Participants) | 7 | 40
  Antepartum Ultrasound, confirmed at delivery | 34.76 (1.24) | 34.68 (1.84)
  Antepartum Ultrasound, not confirmed at delivery: number analyzed (Participants) | 2 | 11
  Antepartum Ultrasound, not confirmed at delivery | 31.50 (2.73) | 34.78 (1.47)
  Antepartum Ultrasound, resolved prior to delivery: number analyzed (Participants) | 0 | 4
  Antepartum Ultrasound, resolved prior to delivery |  | 37.04 (1.55)
  No antepartum diagnosis, Vasa Previa at birth: number analyzed (Participants) | 1 | 1
  No antepartum diagnosis, Vasa Previa at birth | 36.14 (1) | 35.57 (0.4)

ADVERSE EVENTS:
Time Frame: Not applicable to this retrospective study. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: Not applicable to this retrospective study. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Groups:
- Vasa Previa: Women with the diagnosis of Vasa Previa made during the pregnancy or at time of delivery who delivered between January 1, 2000 and December 31, 2012.
  All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Vasa Previa
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes